CLINICAL TRIAL: NCT04749082
Title: Long Term Follow up of Patients With Thoracolumbar Spondylodiscitis Treated Surgically by Posterior Approach in Assiut University Hospitals
Brief Title: Follow up Patients With Thoracolumbar Spondylodiscitis Surgically Treated by Posterior Approach
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Micheal Bassem Elia, Principal investigator, Assiut University
Other Study IDs: spondylodiscitis surgery
Record Dates: First submitted 2021-01-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Spondylodiscitis
Keywords: discitis; Spondylitis; Spine surgery
MeSH Terms: conditions — Discitis; Spondylitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the long term outcomes of patients with thoracolumbar spondylodiscitis treated surgically by posterior approach.

Outcomes include bony fusion, neurological improvement, pain improvement, implant related complication, recurrence of infection and or reoperation rate

DETAILED DESCRIPTION:
spondylodiscitis is characterized by infection that primarily affects the intervertebral disc and adjacent vertebrae. The estimated incidence of spondylodiscitis, ranging from 0.2 to 10 per 100,000 inhabitants per year, has increased in recent years, which is likely associated with an aging population, higher prevalence of chronic disease, and more effective diagnostic techniques. Spondylodiscitis is a life-threatening disease with a mortality rate of 2-20% that is often associated with potential complications, such as paraspinal abscess, epidural abscess, meningitis, spinal instability, and neurologic deficiency. The relapse rates were reported to be as high as 32% in the literature. The aims of this study are to evaluate improvements, complications, recurrence and reoperation rates in Assiut university hospitals.

ELIGIBILITY:
Inclusion Criteria:

* • All patients had thoracolumbar spondylodiscitis from number 1 thoracic vertebra till number 1 sacral vertebra.

  * Treated surgically by posterior approach only.

Exclusion Criteria:

* • Patients with incomplete follow up.

  * Multifocal discitis.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All Patients suffered from thoracolumbar spondylodiscitis and treated surgically by posterior approach in Assiut university hospitals from January 2016 to December 2017
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Bony fusion success | 2 years
  the degree of bridging bone across the fused vertebral bodies by using x-ray, CT scan and MRI if needed

SECONDARY OUTCOMES:
modified Oswestry disability index | 2 years
  for patient quality of life postoperative
visual analogue scale | 2years
  the amount of pain sensed by the patient pre and post-operative
American spinal injury Association (ASIA) Impairment score | 2 years
  to asses neurological outcomes pre operative and at 2 years follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Essam M Abdelmoneim Elmorshidy, Lecturer, Principal Investigator — Assiut University; El Moataz A Zohny El Sabrout, professor, Study Chair — Assiut University; Belal O Mohamed Elnady, Lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Kamal AM, El-Sharkawi MM, El-Sabrout M, Hassan MG. Spondylodiscitis: experience of surgical management of complicated cases after failed antibiotic treatment. SICOT J. 2020;6:5. doi: 10.1051/sicotj/2020002. Epub 2020 Feb 14. PMID 32057290
- [Background] Berbari EF, Kanj SS, Kowalski TJ, Darouiche RO, Widmer AF, Schmitt SK, Hendershot EF, Holtom PD, Huddleston PM 3rd, Petermann GW, Osmon DR, Infectious Diseases Society of America. 2015 Infectious Diseases Society of America (IDSA) Clinical Practice Guidelines for the Diagnosis and Treatment of Native Vertebral Osteomyelitis in Adults. Clin Infect Dis. 2015 Sep 15;61(6):e26-46. doi: 10.1093/cid/civ482. Epub 2015 Jul 29. PMID 26229122
- [Background] El-Sharkawi MM, Said GZ. Instrumented circumferential fusion for tuberculosis of the dorso-lumbar spine. A single or double stage procedure? Int Orthop. 2012 Feb;36(2):315-24. doi: 10.1007/s00264-011-1401-9. Epub 2011 Nov 10. PMID 22072401